CLINICAL TRIAL: NCT04266951
Title: Singstrong: Singing for Better Lung Health
Acronym: Singstrong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NF1
Record Dates: First submitted 2019-06-14; First posted 2020-02-12 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Disease; COPD
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Pilot study: Pre and post intervention with a single patient cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group singing and breathing control training (Other)
  Interventions: Behavioral: Singstrong:

INTERVENTIONS:
Behavioral: Singstrong: — Group singing and breathing control training

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a pervasive, insidious condition associated with catastrophic socioeconomic, healthcare and personal implications. This proposal outlines how a group singing intervention, led by clinical personnel and a community singing leader, can address these challenges. Built upon existing ties between the Principal Investigator (PI) and local COPD support group, this project is co-designed by patients and clinicians. Modelled on similar interventions internationally, this project is pioneering in Ireland. Outputs will include a participant-led symposium and three community COPD choirs, in addition to a number of academic publications. This project is funded by the Irish Research Council (IRC) "New Foundations" scheme.

DETAILED DESCRIPTION:
Brief Background:

Approximately 440,000 Irish people suffer from Chronic Obstructive Pulmonary Disease (COPD) (Health Service Executive (HSE), 2018) and it is the fourth most common cause of death, after lung cancer, heart disease and stroke. In addition to many physical issues, patients lack the physical endurance or confidence to participate fully in their lives, leading to isolation, social exclusion and co-morbid depression and anxiety. Addressing the management of people with COPD was highlighted as an urgent priority in the Government's 2017 National Healthcare Quality Reporting System annual report. This application proposes a community-based singing intervention replicating that successfully delivered by the British Lung Foundation (BLF) (https://www.blf.org.uk/support-for-you/singing-for-lung-health). This project is unique in Ireland, and builds on established ties between the (Principal Investigator) PI and the local COPD community. It is supported by COPD Support Ireland.

Study design:

* This study is a pre-post intervention study involving a cohort of COPD patients who are members of regional COPD support groups in Limerick, Ennis and Nenagh.
* Pre-intervention testing will involve self-reported measures wellness using standardised tools as well as a walking test (6-minute walking test (6MWT) and spirometry to asses lung function.
* The intervention is an eight-week singing intervention led by an experienced singing instructor who will be provided with relevant training on singing with lung impairment. Participants will also be provided with a compact disk (CD) for between intervention practice at their own discretion.
* Post-intervention testing will repeat tests done at baseline. Testing will be carried out in both instances by the PI and clinical staff from the geographical area.

Focus groups will be conducted with a sample from each group to support a qualitative evaluation of the intervention.

Participants:

Approximately 30 participants from each region will be invited to participate. Participants must have a diagnosis of COPD, must be clinically stable, and not have suffered an exacerbation in the 2 weeks prior to testing.

Participants have been sourced through the clinicians involved in this study, and the teaching contacts of the PI.

Procedures/Methods :

Planing stage: April/May 2019

* Community singing leader will attend United Kingdom (UK) training course delivered by BLF "Singing for Lung Health" leaders. - Liaise with three regional COPD patient groups (Limerick, Ennis, Nenagh) to gather informed consent, and finalise intervention details.
* Design and record CD featuring exercises and songs for home practice for participants. These will be provided freely to participants and based on song preference of patient-partners, and informed by disease limiting factors.
* Baseline testing of participants as discussed will take place in a community setting where the groups normally meet for other exercise and social activities.

Intervention stage: June/July 2019

* The intervention will comprise eight weekly one-hour singing sessions. Sessions will be comprised of physical warm-ups, breathing exercises, and vocal exercises such as rhythm and pitch games.
* The intervention will be delivered by the community singing leader and the PI will attend the first session to explain the clinical relevance of exercises.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an existing diagnosis of COPD according to recognised diagnostic criteria, must be clinically stable, and not have suffered an exacerbation in the 2 weeks prior to testing.
* All participants must be at least 18 years of age. There is no upper age limit.
* Participants may be male or female.
* They must have a good command of written and spoken English.

Exclusion Criteria:

* Lack of a clinical diagnosis of COPD
* Presence of physical of psychological co-morbidities precluding participation in either testing or intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Patient anxiety and depression | 8 weeks
  Hospital Anxiety and Depression Scale (HADS). This questionnaire is widely used to measure anxiety and depression in a general medical population of patients. The questionnaire features seven questions for anxiety and seven for depression of which can be answered within 2 - 5 minutes. Each item is scored from 0-3 with a higher score indicating a greater presence of either anxiety or depression. Maximal (worst) score for either factor is 21.
Functional capacity | 8 weeks
  Six minute walk test (6MWT). The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. This is measured in metres with levels of oxygen saturation and heart rate pre and post the test also recorded.
Disease impact | 8 weeks
  COPD Assessment test (CAT). The CAT is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. This is a patient-completed questionnaire assessing all aspects of the impact of COPD (cough, sputum, breathlessness, chest tightness, confidence, activity, sleep and energy levels) There are 8 questions on a 1 to 5 point scale. A higher score indicates more disease impact. Max score is 40.

SECONDARY OUTCOMES:
Lung function | 8 weeks
  Spirometry: The main measures recorded will include FEV1, or forced expiratory volume, is a measurement taken from a pulmonary function test. It calculates the amount of air that a person can force out of their lungs in 1 second.FVC, or Forced Vital Capacity, refers to the total amount of air that a person can exhale, will also be recorded. The ration of FEV1/FVC will also be recorded, as this provided an objective measure of the presence of disease. FEV1/FVC < 0.70). Disease severity in persons below a ratio of 0.7 is indicated by the value of FEV1. Mild FEV1 ≥ 80% predicted, Moderate 50% ≤ FEV1 < 80% predicted, Severe 30% ≤ FEV1 < 50% predicted, Very Severe FEV1 < 30% predicted.
Qualitative evaluation of intervention | 8 weeks
  Focus Groups: Focus group interviews with participants from each of the three choirs will be conducted to establish the effectiveness of the intervention, to establish what went well, and points for improvement in further iterations. Focus groups will be comprised of between 5 and 8 people, with a semi-structured design.

CONTACTS AND LOCATIONS:
Overall Officials: Roisin Cahalan, PhD, Principal Investigator — University of Limerick
Locations (1):
- University of Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: No